CLINICAL TRIAL: NCT03646084
Title: The Impact of a Sleep and Circadian Intervention Program (SCIP) in Chronic Musculoskeletal Pain (CMP) Rehabilitation: a Feasibility PILOT Study
Brief Title: Sleep and Circadian Intervention Program for Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Hospital General Universitario de Guadalajara (Unknown); Hospital Universitario La Paz (Other); Fundación para la Formación y la Investigación de los Profesionales de la Salud- Cáceres (FUNDESALUD) (Unknown); Instituto de Investigación Biomédica de Lleida (Unknown); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, OlgaMediano, Principal Investigator, Consorcio Centro de Investigación Biomédica en Red (CIBER)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIBERES-FES2018-05
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain; Sleep; Circadian Rhythm Disorders
Keywords: pain; sleep; circadian rhythm
MeSH Terms: conditions — Chronic Pain; Chronobiology Disorders; Pain | interventions — Sleep; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Intervention Program (SCIP) (Experimental): Based on the results of the studies, patients will be treated according to current guidelines: 1) Improve rest/activity rhythms. 2) To treat and control Sleep Disorder Breathing. 3) To improve anxiety, depression and insomnia. 4) To treat RLS if needed. 5) To try opioid dose reduction. 6) To trial of non-opioid in lieu of opioids. 7) Avoiding use of benzodiazepines, sedatives, hypnotics. 8) Caution against alcohol use.
  Interventions: Other: Sleep and Circadian Intervention Program (SCIP) plus rehabilitation program
- Control (Active Comparator): Rehabilitation according to current clinical practice.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Sleep and Circadian Intervention Program (SCIP) plus rehabilitation program — To study circadian rhythm disorders and sleep disorders and develops the SCIP to improve sleep in the patients.
  Arms: Sleep Intervention Program (SCIP)
Other: Rehabilitation program — Rehabilitation program current clinical practice
  Arms: Control

SUMMARY:
Musculoskeletal pain has become in a major problem related to its prevalence, treatment cost, absenteeism, quality of life impairment, disability and drugs consumption. The difficulty in musculoskeletal pain control ends in the abuse of drugs by these patients, including opioids. This drugs consumption has become a health problem in the United States and around the world related to their increasing abuse mainly between 2002 and 2011 and has had an impact in the numbers of deaths caused by opioids prescription (reaching 16,651 deaths in United States in 2010). Pain is clearly associated with sleep disturbances (50-80% of these patients suffer from a sleep problem), and in turn poor sleep quality leads to increased pain sensitivity. There is evidence showing that improving sleep disturbance co-occurring pain would improve, and some may reduce the use of opioids in specific patients on long-term opioid therapy. In spite of this reciprocal relationship between sleep and pain only few programs take into account the management of sleep disorders as a non-pharmacological measure for pain control. The hypothesis is: "to address sleep and circadian disorders (SCD) using a Sleep and Circadian Intervention Program (SCIP) in patients treated with rehabilitation by chronic musculoskeletal pain (CMP) optimizes the rehabilitation outcomes and reduces opioids consumption".

Main goal:

The aim of this PILOT study is to evaluate the feasibility of the protocol of the present study that aims to assess the improvement in rehabilitation outcomes and decrease in opioid consumption, through the management of sleep disorders.

Methodology Using a randomised (1:1) controlled feasibility study, 50 men and women will be included to evaluate methodology and identify the potential outcome of the main project. Subjects older than 18 years included in a rehabilitation program by musculoskeletal lumbar pain lasting more than three months will be recruited. Basal Visit (BV): After the signature of informed consent, a medical history, physical exam, evaluation of the pain perception (EQ5D5L), quality of life evaluation (SF36 and FOSQ), mood and anxiety (HADS y PASS20), circadian rhythm study and drugs consumption will be evaluated in both groups. Patients will be randomized to control group (usual rehabilitation program) or intervention group (usual rehabilitation program + sleep circadian intervention program-SCIP). The patient in the SCIP program will received the next intervention: 1) Educational and circadian rhythm intervention: general sleep hygiene recommendation and promotion of daily physical activity. 2) Sleep studies for sleep quality and sleep disorders diagnosis: full polysomnography 3) Sleep questionnaires for another sleep disorders. Based on the results of the studies, patients will be treated according to current guidelines for the management of sleep disorders. 6 month after the SCIP starts patients will be evaluated in the End of Study Visit (EOS) as in the BV and also in their functional improvement and health resources consumption.

DETAILED DESCRIPTION:
Hypothesis: to address sleep and circadian disorders (SCD) using a Sleep and Circadian Intervention Program (SCIP) in patients treated with rehabilitation by chronic musculoskeletal pain (CMP) optimizes the rehabilitation outcomes and reduces opioids consumption.

The Main Objective of this PILOT study is to evaluate the feasibility of the protocol of the present study that aims to assess the improvement in rehabilitation outcomes and decrease in opioid consumption, through the management of sleep disorders.

Secondary objectives of the PILOT study:

1. To identify the primary outcome to evaluate the hypothesis. Evaluate relevance and observed change of the main outcome for the main study. It will allow investigators to evaluate the effect size and variability of the SCIP in the opioids consumption in a sample of our population to determine if this is the potential outcome for the main project.
2. To determine the patient inclusion rhythm (recruitment rate) and, if necessary, the reasons for non-recruitment.
3. To determine the follow-up rate and reasons for loss to follow-up.
4. To test the sleep circadian study's methodology in this type of population.
5. To assess the acceptability, implementation and preliminary efficacy of the SCIP.
6. To evaluate adherence and fidelity to the SCIP through recruitment and retention.
7. To determine the data acquisition rate, amount of missing data and reasons for loss.
8. To evaluate the safety of the program.
9. To characterize the effect observed in the intervention in order to properly calculate the sample size necessary for the main study.

Methodology:

Type of study: This study aims to be the pilot project of a large-scale international randomized controlled trial that will include a total of 1.000 patient internationally. In this pilot study, using a randomised (1:1) feasibility study, 50 patients in a rehabilitation program referred to treatment for CMP lumbar pain will be recruited. The pilot study will have a total duration of 18 months (12 months of recruitment + 6 months follow-up) and all the interventions included in the methodology of the main study will be carried out in the participating patients. As a feasibility trial, aspects of feasibility will be determined and estimates of effect size and measured variability will be calculated to inform future planned study. The data for this study will be collected from standard measures administered in their basal visit (BV), immediately prior to the initiation of the SCIP, and 6 months after the initiation of the program (End of study visit-EOS). Randomisation to allocate participants to either intervention or control group will be performed immediately following the baseline assessment, and intervention delivery (SCIP) will begin directly after the BV. Participants will be then reassessed at 6 months after the baseline (EOS) as in the BV and for functional improvement and health resources consumption. Inclusion criteria: 1) Subjects older than 18 years 2) Inclusion in a rehabilitation program by musculoskeletal lumbar pain lasting more than three months 3) Patients have no severe reading or learning difficulty 4) Signature of informed consent. Exclusion criteria: 1) Severe psychopathological co-morbidity (e.g. the presence of schizophrenia, bipolar disorders…) 2) Co-morbid malignant/terminal diseases (e.g. HIV/AIDS, cancer) 3) Shift-workers and people who work making transmeridian travels.

All patients will provide written consent for their data to be used in an anonymized form for research purposes and project will have ethics and research and development committee approval prior to the start.

Basal Visit: All participants will be asked to provide in the BV the basic demographic information, medical characteristics (age, gender, job, medication), pain characteristics (pain cause, time, location and intensity) and a basic physical exam (blood pressure, height, weight, neck, hip and waist circumference), a drugs test will be performed to assess opioids consumption and a circadian rhythm study (individual activity rhythms will be measured noninvasively with Kronowise® [with European Community marking for this indication] in all patients). To evaluate the effect of the SCIP pain reduction may not be sufficient for a comprehensive evaluation of the overall benefit of the intervention. The complexity of chronic pain and its negative impact on diverse aspects of function should be evaluated: 1a. To evaluate the improvement of pain perception and pain intensity control: pain intensity, sensory pain ratings and affective pain ratings will be measured before and after the intervention in both groups. To provide this multidimensional assessment of pain the 5-level EQ-5D version (EQ-5D-5L) will be completed in basal visit and after intervention.1b. To evaluate the improvement in quality of life (QoL) measured it will be measured by QoL questionnaires (SF36 and FOSQ) before and after the intervention and 1c. To measure the improvement in mood and anxiety patients will answer the Hospital Anxiety and Depression Scale (HADS) and Pain Anxiety Symptoms (Scale-PASS20).

Groups: The patients will be selected by their rehabilitation doctor who will establish the indication and dose of the necessary medication to control the pain, according to the criteria of conventional clinical practice.

Patients will be randomized to:

1 Control group. Rehabilitation according to current clinical practice. 2 SCIP group. Rehabilitation according to current clinical practice + specific actions in the treatment group (the next action in this point 2 will be undergo only in the SCIP group): 2a. Educational and circadian rhythm intervention: 2a. I - General sleep hygiene recommendations. 2a. II - Promotion of daily physical activity: determine sleep circadian patterns during rehabilitation: Each participant will record his/her sleep periods in a sleep log. In addition, individual rest/activity, distal skin temperature and light exposure rhythms will be measured noninvasively with a watch-like device (Kronowise ®) during 7 consecutive days and nights. Sleep disturbances as sleep onset latency longer than 30 minutes, more than two waking episodes per night, total sleep time shorter than 6.5 hours or a sleep efficiency lower than 85% will be take into account and submitted to the specialist if necessary. Specific circadian habits modification advise or treatment will be given depending in the results. All this information will be collected and analysed to determine sleep and circadian hygiene and the circadian rhythms of the above-mentioned variables in the BV and after the SCIP (EOS).

2b. Describe the sleep disorders related to chronic pain by applying sleep studies to evaluate sleep quality and to diagnose sleep disturbances during rehabilitation: full Polysomnography 2c. Describe other sleep disorders by applying specific questionnaires: To evaluate quality of sleep the Pittsburgh questionnaire will be performed, the Epworth Sleepiness scale to assess daytime hypersomnolence and to diagnose other sleep disorders such as insomnia and restless legs syndrome (RLS) the Insomnia Severity Index (ISI) and the RLS criteria will completed respectively.

2d. Therapeutic intervention related to the results obtained in the mentioned studies (2 a, b and c): advice/treatment will be recommended to determine the effect of the specific interventions decided (pharmacological or non-pharmacological) related to SCD detected in 2 a,b and c. Based on the results of the studies, patients will be treated according to current guidelines for the management of sleep disorders and taking into account the following recommendations: 1) Interventions that improve rest/activity rhythms: Sleep Hygiene, bright light therapy and noise control, time of exercise and feeding. 2) To treat and control Sleep Disorder Breathing (including adaptive servo-ventilation and bi-level positive airway pressure ventilation for Central Sleep Apnea if needed). 3) To improve anxiety, depression and insomnia (to apply bright light therapy and refer to a specialist if needed). 4) To treat Legs Restless Syndrome if needed. 5) To try opioid dose reduction. 6) To trial of non-opioid therapies (NSAIDs, antiepileptic drugs, physical therapy, antidepressants…) in lieu of opioids. 7) Avoiding use of benzodiazepines, sedatives, hypnotics. 8) Caution against alcohol use.

Blood samples extraction will be obtained from all participants at the beginning of rehabilitation and at the end of follow-up to study to measure serum levels of inflammatory and oxidative stress biomarkers implicated in pain control.

EOS visit: After 6 months of the initiation of the SCIP the BV measurements will be repeated and also an evaluation of the functional improvement and consumption of health resources. The impact of the SCIP will be evaluated in the next aspects: 1a. Improvement of pain perception and pain intensity control. 1b. Improvement in quality of life (QoL). 1c. Improvement in mood and anxiety. 1d. Physical functioning improvement: activity registers from Kronowise ® will be used to assess the physical activity rhythm improvement (specific measures of the affected musculoskeletal component). 1e. Consumption of health resources (pharmacological and non-pharmacological): Pharmacological consumption: Patient pharmacologic sleep and pain agents and dosing will be recorder at basal visit and after the sleep intervention: opioid analgesics, benzodiazepine receptor agonists, nonbenzodiazepine benzodiazepine receptor agonists, melatonin receptor agonists, antidepressants, antipsychotics, anticonvulsants, general analgesic and antihistaminic drugs. Non-pharmacological consumption: days of rehabilitation treatment, visits to emergency department, hospitalization related to pain or CP treatment, duration of sick leave (days of work absenteeism). 1f. Improvement of the circadian system parameters.

Ethics and Safety: There are no expected serious adverse events (SAEs) in this study. The proposed procedures carry minimal risk to participants, and their care and comfort will be ensured throughout. This research will be performed in accordance with the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) standards. Research Ethics Service ethical approval will be sought and confirmed before the start of the trial. The study will be overseen by a steering committee who will act as the data-monitoring committee to consider adverse effects and/or lack of adherence to the protocol.

Sample Size: As this was a feasibility study, a sample size calculation was not performed. The study aimed to recruit 50 patients randomized (1:1) to control group (usual rehabilitation and circadian rhythm study) or intervention group (usual rehabilitation program + sleep circadian intervention program-SCIP) in patients under rehabilitation treatment by musculoskeletal chronic pain on the opioids consumption. Data from key outcome measures were later used to determine the sample size for a definitive trial.

Statistical analysis: Descriptive statistics of mean (standard deviation) or median [interquartile range (IQR)] were estimated for quantitative variables with a normal or non-normal distribution, respectively, while absolute and relative frequencies were used for qualitative variables. Normal distribution was analysed using the Shapiro-Wilks test. Participant characteristics were compared using Student's test, analysis of variance (ANOVA), or non-parametric Mann-Whitney and Kruskal-Wallis tests for non-normal distribution. The statistical level of significance was fixed at 0.05. All analyses were performed using R statistical software, version 3.4.2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years
* Inclusion in a rehabilitation program by lumbar musculoskeletal pain lasting more than three months
* Patients have no severe reading or learning difficulty
* Signature of informed consent.

Exclusion Criteria:

* Severe psychopathological co-morbidity (e.g. the presence of schizophrenia, bipolar disorders…)
* Co-morbid malignant/terminal diseases (e.g. HIV/AIDS, cancer)
* Shift-workers and people who work making transmeridian travels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumed dose | 12 months
  Quantification of decrease dose opioids consumption related through the management of sleep disorders.

SECONDARY OUTCOMES:
Opioids urine drugs test to assess opioids consumption | 12 months
  Quantification of decrease in number of patients with opioids consumption (urine levels) through the management of sleep disorders.
Determine inclusion rhythm. | 6 months
  To determine the patient inclusion rhythm (recruitment rate) and, if necessary, the reasons for non-recruitment.
Number of patients lost in follow up. | 12 months
  To determine the follow-up rate.
Sleep circadian study's methodology | 12 months
  To test the sleep circadian study's methodology in this type of population.
Number of patients that complete the SCIP | 12 months
  To assess the acceptability, implementation and preliminary efficacy of the SCIP.
Number of patients the developed the EOS visit | 12 months
  To evaluate adherence and fidelity to the SCIP through recruitment and retention.
Determine data acquisition. | 18 months
  To determine the data acquisition rate, amount of missing data and reasons for loss.
Number of participants with SCIP-related adverse events as assessed | 12 months
  To evaluate the safety of the program.
Number of patients needed related to the SCIP effect size. | 12 months
  To characterize the effect observed in our intervention in order to properly calculate the sample size necessary for the main study. Data from key outcome measures were later used to determine the sample size for a definitive trial.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Mediano, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)
Locations (1):
- Hospital Universitario de Guadalajara, Guadalajara, Spain

IPD SHARING:
Plan to Share IPD: Undecided